CLINICAL TRIAL: NCT05709574
Title: An Open-Label, Phase II Single-Arm, Window Trial of Tadalafil Effect + Chemotherapy in Patients With Resectable Gastric/GEJ Adenocarcinoma
Brief Title: Tadalafil Effect + Chemotherapy in Resectable Gastric/GEJ Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001728
Record Dates: First submitted 2022-12-15; First posted 2023-02-02 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: PDE5,6i inhibitor; chemotherapeutic cell death; resectable Gastric/GEJ cancer; tadalafil; FLOT chemotherapy; Myeloid Derived Suppressor Cells (MDSCs)
MeSH Terms: interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tadalafil + chemotherapy (Experimental): Subjects will receive Tadalafil monotherapy for 2 weeks followed by Tadalafil in combination with neoadjuvant FLOT chemotherapy for 8 weeks in the window between their cancer diagnosis and surgical intervention.
  Interventions: Drug: Tadalafil 20 MG

INTERVENTIONS:
Drug: Tadalafil 20 MG — Tadalafil 20 mg tablets will be taken daily for 2 weeks alone and then for 8 weeks in combination with neoadjuvant chemotherapy in the window between gastric/GEJ adenocarcinoma diagnosis and interventional surgery.
  Other Names: Cialis

SUMMARY:
The goal of this clinical trial is to assess the ability of Tadalafil alone and in combination with neoadjuvant FLOT (5-Fluorouracil, Oxaliplatin, and Docetaxel) chemotherapy to suppress myeloid derived suppressor cells (MDSCs) in patients with resectable gastric or gastroesophageal junction adenocarcinoma. Resectable means the tumor may be removed through surgical intervention. Neoadjuvant chemotherapy is chemotherapy received before the primary course of treatment i.e.surgical intervention.

The main questions it aims to answer are:

* Is Tadalafil treatment with FLOT feasible and safe?
* How does tadalafil treatment with FLOT affect the tumor microenvironment (TME)?
* Will 8 weeks of neoadjuvant exposure to tadalafil with chemotherapy reduce MDSCs in the TME?

Participants will receive Tadalafil for 14 days followed by combination of Tadalafil + FLOT for approximately 8 weeks as a part of standard of care neoadjuvant treatment in the window between cancer diagnosis and surgical intervention to remove their tumor. Tumor tissue, blood, and urine will be collected at the start of the study, after 2 weeks of treatment with Tadalafil alone, and around the time of surgical intervention. Saliva will also be collected at the start of the study.

DETAILED DESCRIPTION:
Despite the availability of multimodality approaches for localized gastric cancer, the survival rates remain dismal for resectable disease. There is a large unmet need to identify new therapeutic options, to be used in combination with chemotherapy and to improve survival outcomes. Emerging data have shown the implication of myeloid derived suppressor cells (MDSCs) in the alteration of tumor microenvironment. The MDSCs are involved in tumor progression by promoting immune suppression, tumor angiogenesis, drug resistance, tumor metastasis and limiting the effects of cancer immunotherapy. In vitro and animal studies have demonstrated that phosphodiesterase 5 inhibitors (PDE5i) such as Sildenafil or Tadalafil inhibit MDSCs, augment the endogenous antitumor immunity and improve the effectiveness of chemotherapy. There have been similar reports of enhanced chemotherapeutic efficacy with PDE5i in murine models of melanoma, multiple myeloma, lung, breast, head and neck, colorectal and brain cancer. PDE5 inhibitors suppress nitric oxide synthetase (Nos)-expressing myeloid derived stem cells (MDSCs). There have been no prior clinical studies using a PDE5,6 inhibitor to enhance chemotherapeutic cell death in the upper gastrointestinal cancers. Therefore, the investigators propose this trial to study the effect of the long-acting PDE5,6i Tadalafil in combination with chemotherapy (FLOT) in resectable Gastric/GEJ cancers.

This is a single arm, phase II, window trial to assess the ability of Tadalafil to suppress MDSCs as monotherapy and in combination with neoadjuvant FLOT chemotherapy in patients with resectable gastric or gastroesophageal junction adenocarcinoma.

The study will enroll 10 patients. Patients will receive Tadalafil for 14 days followed by combination of Tadalafil + FLOT for approximately 8 weeks as a part of standard of care neoadjuvant treatment. Tumor specimens, blood, and urine will be collected at baseline, after 2 weeks of monotherapy treatment with Tadalafil, and around the time of surgical intervention to analyze the tumor microenvironment (TME) and to determine whether PDE5, 6 inhibition reduces the immune suppressive microenvironment. Saliva will also be collected at baseline.

Hypothesis: The investigators hypothesize that daily dosing of Tadalafil with chemotherapy will significantly reduce myeloid-derived suppressor cells (MDSCs) in the TME.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I-III (T1-3Nx) Gastric or GEJ (Siewert 3) adenocarcinoma, confirmed by histology or cytology.
2. Radiographically measurable disease by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Images (MRI or CT scan) must be completed within 28 days prior to treatment start.
3. Age ≥ 18 years.
4. Adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 14 days before first dose of study treatment:

   1. Absolute neutrophil count (ANC) ≥ 1500/µL without granulocyte colony-stimulating factor support within 2 weeks.
   2. White blood cell count ≥ 2500/µL including Lymphocyte count ≥ to 500/µL.
   3. Platelets ≥ 100,000/µL without transfusion.
   4. Hemoglobin ≥ 9 g/dL (≥ 90 g/L).
   5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN) with the following exceptions: Patients with documented liver metastases: AST and ALT ≤ 5 x ULN. Patients with documented liver or bone metastases: ALP ≤ 5 x ULN.
   6. Total bilirubin ≤ 1.5 x ULN (for subjects with Gilbert's disease ≤ 3 x ULN).
   7. Serum albumin ≥ 2.8 g/dl.
   8. (PT)/INR or partial thromboplastin time (PTT) test < 1.3 x the laboratory ULN.
   9. Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 40 mL/min using the Cockcroft- Gault equation:

      * Males: (140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)
      * Females: [(140 - age) x weight (kg)/(serum creatinine [mg/dL] × 72)] × 0.85
5. ECOG performance status ≤ 1.
6. Sexually active fertile subjects and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 6 months after the last dose of study treatment.
7. Female subjects of childbearing potential must not be pregnant at screening. Female subjects are considered to be of childbearing potential unless one of the following criteria are met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. Note: Documentation may include review of medical records, medical examinations, or medical history interview by study site.
8. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Prior treatment for gastric cancer.
2. Prior treatment with Tadalafil or other PDE inhibitors within 28 days.
3. Known metastatic disease.
4. The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

   a) Cardiovascular disorders: i. Congestive heart failure New York Heart Association Class II-IV, unstable angina pectoris, serious cardiac arrhythmias.

   ii. Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment. iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose of study treatment. iv. Subjects with a diagnosis of incidental, subsegmental PE or DVT within 6 months are allowed if stable, asymptomatic, and treated with a stable dose of permitted anticoagulation (see exclusion criterion #6) for at least 1 week before first dose of study treatment. v. Ventricular tachyarrhythmia requiring ongoing treatment vi. Unstable angina pectoris vii. Sinus bradycardia b) Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: i. The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction. ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose of study treatment. iii. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.
5. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis (see Appendix III for a more comprehensive list of autoimmune diseases and immune deficiencies), with the following exceptions:

   1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
   2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met: i. Rash must cover < 10% of body surface area. ii. Disease is well controlled at baseline and requires only low-potency topical corticosteroids.

   iii. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
6. Active infection requiring systemic treatment with the following exceptions:

   1. Urinary tract infections.
   2. HCV on active treatment.
7. Patients with SARS-COV-2 infections with the following exceptions:

   a) Recovery from active symptoms 30 days prior to treatment start.
8. Known history of infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or a known positive test for tuberculosis due to tuberculosis infection.
9. Concomitant medication uses of nitrates, α-blockers and other interacting medications (CYP3A4 inhibitors and CYP3A4 inductors).
10. Other clinically significant disorders as deemed by the investigator, that would preclude safe study participation.

    1. Serious non-healing wound/ulcer/bone fracture.
    2. Uncompensated/symptomatic hypothyroidism.
    3. Moderate to severe hepatic impairment.
11. Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Subjects must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
12. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    1. Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained.
    2. Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
13. Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment of within 6 months after the final dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result within screening. Test will need to be repeated if last completed >3 days prior to initiation of study treatment.
14. Inability to swallow tablets.
15. Previously identified allergy or hypersensitivity to components of the study treatment formulations.
16. Previous episode of Non-arteritic anterior ischemic optic neuropathy (NAION)
17. Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluating the safety and tolerability of tadalafil treatment with FLOT chemotherapy by assessing the number of participants with treatment related adverse events usting CTCAE v. 5.0. | 10 weeks
  To evaluate the safety and tolerability by assessing the number of participants with treatment related adverse events using CTCAE v5.0.

SECONDARY OUTCOMES:
Pathological response after PDE5 inhibition and treatment using Becker's Criteria | 10 weeks
  To evaluate the pathologic response using Becker's Criteria.
Radiographic response after PDE5 inhibition and treatment based on RECIST1.1 | 10 weeks
  To evaluate the radiologic response based on response evaluation criteria in solid tumors version 1.1 (RECIST1.1)

OTHER OUTCOMES:
Effect of Tadalafil on the myeloid derived suppressor cells (MDSCs) population as measured by 50% change in MDSCs | 8 weeks
  To evaluate the effect of Tadalafil on the MDSC population in patients with operable, Gastric/GEJ adenocarcinoma as measured by 50% change in MDSCs following approximately 8 weeks of neoadjuvant exposure.
Change in tumor-intrinsic genetic biomarkers TLR9 SNP rs5743836 before and after treatment. | 10 weeks
  To evaluate tumor-intrinsic genetic biomarkers TLR9 SNP rs5743836 before and after treatment.
Change in intrinsic genetic biomarker MIR130b before and after treatment. | 10 weeks
  To evaluate intrinsic genetic biomarker MIR130b before and after treatment.
Change in tumor activation markers, NFkB, before and after treatment. | 10 weeks
  To evaluate tumor activation markers such as NFκB before and after treatment.
Change in intrinsic genetic biomarker SLFN12L before and after treatment | 10 weeks
  To evaluate intrinsic genetic biomarker SLFN12L before and after treatment.
Change in intrinsic genetic biomarker cGMP before and after treatment. | 10 weeks
  To evaluate intrinsic genetic biomarker cGMP before and after treatment.
Change in tumor tissue markers of tumor differentiation, TFF2, before and after treatment. | 10 weeks
  To evaluate markers of tumor differentiation TFF2 before and after treatment.
Change in markers of tumor differentiation CDX2 before and after treatment. | 10 weeks
  To evaluate markers of tumor differentiation CDX2 before and after treatment.
Change in markers of tumor proliferation Ki67 before and after treatment. | 10 weeks
  To evaluate markers of tumor proliferation Ki67 before and after treatment.
Change in plasma biomarker MIR130b before and after treatment. | 10 weeks
  To evaluate plasma biomarker MIR130b before and after treatment.
Change in urine biomarker MIR130b before and after treatment. | 10 weeks
  To evaluate urine biomarker MIR130b before and after treatment.
Change in PBMCs biomarkers MIR130b before and after treatment. | 10 weeks
  To evaluate PBMCs biomarkers MIR130b before and after treatment.
Change in PBMCs biomarkers SLFN12L before and after treatment. | 10 weeks
  To evaluate PBMCs biomarkers SLFN12L before and after treatment.
Change in saliva biomarker TLR9 SNP expression. | Saliva will be collected at baseline
  To evaluate saliva biomarker TLR9 SNP expression.

CONTACTS AND LOCATIONS:
Overall Officials: Junaid Arshad, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center at UMC North/University Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No